CLINICAL TRIAL: NCT07290660
Title: Effectiveness of Graded Motor Imagery and Task-Oriented Exercise Training in Shoulder Impingement Syndrome
Brief Title: Graded Motor Imagery and Task-Oriented Exercise in Shoulder Impingement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Yeliz ÇIRAK, Principal Investigator, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FBU
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Shoulder Impingement Syndrome; Pain; Motor Imagery Training; Task Oriented Training
Keywords: Shoulder impingement syndrome; Graded motor imagery; Task-oriented exercise; Rehabilitation; pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain | interventions — Electric Stimulation Therapy

STUDY DESIGN:
Intervention Model Description: This study uses a three-arm parallel-group design. Participants will be randomly assigned to one of three groups: conventional physiotherapy, graded motor imagery, or task-oriented exercise training. All groups will receive a 6-week intervention without crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Conventional Physiotherapy (Active Comparator): Participants in this group will receive conventional physiotherapy, including standardized electrotherapy and routine therapeutic exercises for shoulder impingement syndrome, for 6 weeks
  Interventions: Other: Electrotherapy + Conventional Exercise Group
- Graded Motor Imagery (Active Comparator): Participants in this group will receive a 6-week graded motor imagery program in addition to standardized electrotherapy
  Interventions: Other: Electrotherapy + Conventional Exercise Group; Other: The graded motor imagery program
- Task-Oriented Exercise Training (Active Comparator): Participants in this group will receive a 6-week task-oriented exercise training program in addition to standardized electrotherapy.
  Interventions: Other: Electrotherapy + Conventional Exercise Group; Other: The task-oriented exercise program

INTERVENTIONS:
Other: Electrotherapy + Conventional Exercise Group — All participants will receive an electrotherapy program consisting of TENS (100 Hz, 20 minutes), ultrasound (1.5 W/cm², 6 minutes), and cold pack application (15 minutes), delivered 5 days per week for 6 weeks. The conventional exercise program includes wand exercises (flexion, abduction, extension, external/internal rotation), Codman exercises in multiple directions, and finger ladder exercises with a 5-second hold at end range. Strengthening exercises will be performed without resistance during the first week, followed by progressive TheraBand® resistance from week two. Posterior, anterior, and inferior capsule stretching, pectoral stretching, and shoulder-scapular mobilization will be performed under physiotherapist supervision. Exercises will be applied twice weekly for 6 weeks, with 3 sets of 10 repetitions.
Other: The graded motor imagery program — The graded motor imagery program consists of 2 weeks of laterality training, 2 weeks of motor imagery, and 2 weeks of mirror therapy. Laterality training will be performed using the Recognise™ Shoulder app (NOI), where participants identify whether presented images show a right or left shoulder. Training will be conducted twice weekly for 2 weeks. Motor imagery includes viewing shoulder movement images (flexion 180°, abduction 180°, external rotation 90°, internal rotation 90°, extension 45°) and mentally rehearsing the movements for 3 sets of 10 repetitions. Mirror therapy requires participants to view the reflection of their unaffected shoulder and perform the imagined movements. Mirror therapy will also be applied twice weekly for 2 weeks, with 3 sets of 10 repetitions
  Arms: Graded Motor Imagery
Other: The task-oriented exercise program — The task-oriented exercise program is based on daily activities related to DASH and SPADI items, focusing on functional shoulder movements including flexion, abduction, extension, and rotation. Exercises will be performed twice weekly for 6 weeks, 3 sets of 10 repetitions. Weeks 0-2 include placing an object on a front shelf, placing an object on a side shelf, placing the hand on the back, touching the neck, washing a plate, and wiping a wall within pain limits. Weeks 2-4 include changing an overhead light bulb, washing hair, combing hair, putting on and taking off a pullover shirt, and donning a jacket or cardigan. Weeks 4-6 include placing a 0.5-kg weight on an overhead shelf (front and side), washing or scratching the upper and lower back, and placing a wallet in the back pocket.
  Arms: Task-Oriented Exercise Training

SUMMARY:
This study aims to compare the effects of graded motor imagery and task-oriented exercise training in individuals with shoulder impingement syndrome. A total of 66 participants aged 25-65 years will be randomly assigned to one of three groups: conventional physiotherapy, graded motor imagery, or task-oriented exercise training. All groups will receive standardized electrotherapy, while the intervention groups will additionally complete 6-week graded motor imagery or task-oriented exercise programs.

Primary outcomes include pain intensity, shoulder range of motion, muscle strength, proprioception, functional status, kinesiophobia, laterality recognition, movement imagery ability, and patient satisfaction. Assessments will be conducted before and after the intervention by the same physiotherapist. The study aims to determine whether motor imagery-based or task-oriented rehabilitation provides additional benefits compared with conventional physiotherapy in individuals with shoulder impingement syndrome.

DETAILED DESCRIPTION:
This study investigates the effects of graded motor imagery (GMI) and task-oriented exercise training on individuals diagnosed with shoulder impingement syndrome. Shoulder impingement is a common musculoskeletal problem that leads to pain, restricted mobility, reduced muscle strength, proprioceptive deficits, and functional limitations. Conventional physiotherapy approaches may not always be sufficient to address the complex sensorimotor deficits associated with this condition. Therefore, this study aims to evaluate whether GMI or task-oriented exercise programs can provide additional therapeutic benefits beyond standard physiotherapy.

A total of 66 participants, aged 25 to 65 years, who meet the diagnostic criteria for shoulder impingement syndrome, will be included. Participants will be randomly assigned to one of three groups:

Conventional physiotherapy (control group)

Graded motor imagery training

Task-oriented exercise training

All groups will receive standardized electrotherapy interventions as part of routine physiotherapy. In addition to this standard treatment, the two intervention groups will engage in a 6-week structured program based on either GMI or task-oriented exercises, depending on group allocation.

Outcome measures will include pain intensity, shoulder range of motion, muscle strength, proprioception, functional level, kinesiophobia, laterality recognition, movement imagery ability, and patient satisfaction. All assessments will be conducted before and after the 6-week intervention by the same physiotherapist to ensure consistency.

The purpose of this study is to determine whether GMI or task-oriented exercise training offers superior improvements in pain, motor performance, proprioceptive control, and functional outcomes when compared with conventional physiotherapy alone. The findings are expected to contribute to evidence-based rehabilitation practices and provide clinicians with additional strategies for managing shoulder impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:Adults aged 25-65 years

Diagnosed with Stage I or Stage II shoulder impingement syndrome by an Orthopedics or Physical Medicine and Rehabilitation physician

Positive Neer and Hawkins tests

Unilateral shoulder pain for at least 3 months

No participation in any physiotherapy program for shoulder problems within the last year

Ability to cooperate and follow instructions

A score of 24 or above on the Standardized Mini-Mental Test -

Exclusion Criteria:

History of previous shoulder surgery

Local corticosteroid injection within the last three months

Presence of uncontrolled neurological, cardiac, or systemic diseases that may interfere with function

Cognitive impairments that may affect proper understanding or execution of the motor imagery program

A score below 24 on the Standardized Mini-Mental Test

-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of Muscle Strength | At baseline and at the end of the 6-week intervention period
  Muscle strength will be assessed using the Lafayette Manual Muscle Tester (MMT). Shoulder flexion, extension, abduction, internal rotation, and external rotation muscle strengths will be evaluated. Three consecutive measurements will be taken for each movement, and the mean value will be recorded.
Assessment of Pain Intensity | At baseline and at the end of the 6-week intervention period
  Pain intensity will be assessed using a 10 cm Visual Analog Scale (VAS), ranging from '0' (no pain) to '10' (unbearable pain). Participants will rate their pain levels before and after the intervention in three conditions: at rest, during activity, and at night
Assessment of Pain Threshold | At baseline and at the end of the 6-week intervention period
  The pain threshold will be assessed using an algometer, a device that measures the pressure at which pain is first perceived. During the measurement, the participant must remain in a relaxed position, and the tip of the algometer must be applied at a 90-degree angle to the tissue. As pressure gradually increases, the participant will be instructed to indicate the moment when pain or discomfort is first felt. This point will be recorded as the pain threshold . In this study, the Commander Echo Algometer will be used to assess pain thresholds. Measurements will be taken from the deltoid muscle, supraspinatus muscle, infraspinatus muscle, and the participant's self-reported most painful area. Each measurement will be repeated three times, and the mean value will be recorded.
Assessment of Shoulder Range of Motion | At baseline and at the end of the 6-week intervention period
  Shoulder range of motion will be assessed using a Baseline goniometer (RMS UK Ltd., Nailsea). The joint movements to be evaluated include flexion, extension, abduction, internal rotation, and external rotation, and the results will be recorded in degrees. For each movement, three consecutive measurements will be taken, and the mean value will be used for analysis
Assessment of Active Joint Position Sense | At baseline and at the end of the 6-week intervention period
  Active shoulder joint position sense will be assessed using a smartphone goniometer application with proven validity and reliability. Elevation angles of 40° and 100° in the scapular plane will be tested. A smartphone will be placed in an armband positioned over the biceps brachii on the tested side. With eyes open, participants will first learn the target angle through passive movement. Then, with eyes closed, the shoulder will be passively positioned at the target angle three times for familiarization. Participants will then actively reproduce the angle. The test will be repeated six times with 5 seconds of rest between trials. The same procedure will be performed for both 40° and 100° elevations on both shoulders.
Assessment of Upper Extremity Function | At baseline and at the end of the 6-week intervention period
  Functional assessment of the shoulder will be performed using the Shoulder Pain and Disability Index (SPADI). SPADI consists of 13 items divided into two subscales: pain and disability. The pain subscale includes five questions related to shoulder pain during activities, while the disability subscale includes eight questions evaluating difficulty in performing daily activities. Both subscale scores and the total score range from 0 to 100, with higher scores indicating greater pain and disability

SECONDARY OUTCOMES:
Assessment of Laterality Recognition | At baseline and at the end of the 6-week intervention period
  Shoulder laterality performance will be assessed using the 'Recognise™' application developed by the Neuro Orthopaedic Institute. The 'Recognise™ Shoulder' section of the app, specifically the 'Vanilla' mode, will be used. A total of 20 shoulder images will be presented for 5 seconds each. Participants will be asked to identify as quickly and accurately as possible whether the displayed image represents a right or left shoulder by pressing the corresponding button on the screen. The percentage of correct responses and reaction time will be recorded as outcome measures.
Assessment of Movement Imagery Ability | At baseline and at the end of the 6-week intervention period
  Movement imagery ability will be assessed using the Movement Imagery Questionnaire-3 (MIQ-3). The questionnaire consists of 12 items. Participants are asked to imagine four different movements using internal visual imagery, external visual imagery, and kinesthetic imagery. They rate the clarity or ease of imagining each movement on a 7-point ordinal scale (1 = very hard to feel/see, 7 = very easy to feel/see)
Assessment of Kinesiophobia | At baseline and at the end of the 6-week intervention period
  Kinesiophobia will be assessed using the Tampa Scale for Kinesiophobia (TSK), developed by Miller, Kori, and Todd. The scale consists of 17 items evaluating fear of injury, reinjury, fear-avoidance beliefs, and activity-related concerns. Each item is scored on a 4-point Likert scale ranging from 1 (strongly disagree) to 4 (strongly agree). Higher scores indicate a higher level of kinesiophobia.
Assessment of Patient Satisfaction | It will be assessed at the end of the 6-week treatment period.
  Patient satisfaction with treatment will be assessed using the Global Rating of Change (GRC) Scale. This scale is widely used in clinical research, particularly in musculoskeletal conditions. It is designed to measure a patient's perceived improvement or deterioration over time, either to determine the effectiveness of an intervention or to track clinical progress. The version used in this study consists of 5 levels and is scored between -2 and +2.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Institute of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No